CLINICAL TRIAL: NCT01117896
Title: Effect of Rescuer Fatigue on Chest Compression Effectiveness
Brief Title: CPR Rescuer Fatigue on Chest Compression Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-5-5367
Record Dates: First submitted 2010-05-04; First posted 2010-05-06 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Rescuer Fatigue During CPR
Keywords: CPR; Rescuer fatigue; Chest Compression effectiveness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adult vs Pedi manikin CC quality (Experimental): The primary objective is to determine whether chest compression deterioration occurs at the same rate in pediatric and adult manikins. The primary endpoint will be the difference in mean number of effective compressions per minute in each manikin at times 1, 2, 5 and 10 minutes.
  Another objective is to identify the correlation between the anaerobic threshold and the deterioration of compressions in each manikin. The endpoint will be the difference between mean time to ineffective compressions (defined as 10 consecutive compressions that fail to meet AHA guidelines for depth and rate) and mean time to anaerobic threshold in each manikin.
  Interventions: Other: Chest compression on adult and pedi manikins
- Stepstool use (Experimental): A third main objective is to determine the effect of the stepstool use on the quality of chest compressions and metabolic demand. The endpoint will be the difference between mean time to ineffective compressions (defined as 10 consecutive compressions that fail to meet AHA guidelines for depth and rate) and mean time to anaerobic threshold in each experimental group.
  Interventions: Other: Use of stepstool during chest compressions

INTERVENTIONS:
Other: Chest compression on adult and pedi manikins — Each participant will be required to perform chest compressions on all 2 manikins, one on each of 2 assigned days. Participants will be randomized to one of 2 groups differing only in the order of manikins compressed, i.e. pediatric-adult; adult-pediatric, etc.
  Other Names: chest compression on adult manikins; chest compression on pedi manikins
  Arms: Adult vs Pedi manikin CC quality
Other: Use of stepstool during chest compressions — In the additional arm of the study, a new cohort of participants will use only the adult manikin on two separate sessions. Participants will be randomized to one of two groups differing only in the use of a stepstool.
  Other Names: chest compression adult manikin
  Arms: Stepstool use

SUMMARY:
This prospective, randomized experimental trial to determine whether the quality of healthcare provider/rescuer chest compressions (CC) deteriorates at the same rate in pediatric models as compared to adult models. To determine the relationship between physiologic/metabolic markers of work in rescuers and chest compression deterioration, and to determine the effect of stepstool use on the quality of chest compressions and metabolic demand. To determine whether the quality of chest compressions deteriorates at the same rate in participants using a stepstool compared to those not using a stepstool.

DETAILED DESCRIPTION:
Context:

Pediatric cardiac arrests result in poor outcomes. Effective chest compressions improve survival in such patients. Unfortunately, compressions are generally inadequately performed and the quality of compressions given deteriorates rapidly with time. Current American Heart Association (AHA) guidelines call for faster and deeper chest compressions with minimization of interruptions. The effect of fatigue on operational performance while adhering strictly to these AHA guidelines is unknown. In addition, there is little pediatric data on rescuer fatigue and chest compression deterioration. Also, the use of a stepstool may affect the quality of chest compressions and may also have an impact on the fatigue of the rescuer. Understanding the biomechanics during optimal chest compression performance may prove useful in the recommendations of conditions and equipment for execution of more effective chest compressions during a cardiac arrest. We will aim to observe and understand the biomechanical qualities that allow for the most effective compressions.

Objectives:

1. To determine whether the quality of chest compressions deteriorates at the same rate in pediatric models as compared to adult models. To determine the relationship between physiologic/metabolic markers of work in rescuers and chest compression deterioration.
2. To determine the effect of stepstool use on the quality of chest compressions and metabolic demand. To determine whether the quality of chest compressions deteriorates at the same rate in participants using a stepstool compared to those not using a stepstool.

Study Design/Setting/Participants:

This prospective, randomized experimental trial will be performed at the Children's Hospital of Philadelphia. Participants will be healthcare practitioners who routinely provide chest compressions in the course of their work. Lay practitioners will be excluded.

Study Measures:

Participants will be asked to perform continuous chest compressions on pediatric and adult sized manikins. Compression rate, depth, applied force as well as participant physiologic work efficiency and anaerobic threshold will be recorded. To evaluate the second objective, a new cohort of participants will perform continuous chest compressions on an adult sized manikin with and without a stepstool.. Compression rate, depth, applied force as well as participant physiologic work efficiency and anaerobic threshold will also be recorded. Videotaping of each subject will also be used for comparison of subjective assessment of chest compression quality and objective chest compression quality data.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 22 to 65 years.
2. Resident physicians, fellows, attendings, nurses and emergency medical technicians (EMTs) who routinely perform chest compressions in the Critical Care units and Emergency Department.

Exclusion Criteria:

1. Lay practitioners
2. Pregnant women
3. Chronic medical Condition limiting exertional capacity

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Compression Quality | 2 years
  The primary endpoint will be the difference in mean number of effective compressions per minute in each manikin at times 1, 2, 5 and 10 minutes.
Metabolic expenditure | 2 years
  The endpoint will be the difference between mean time to ineffective compressions (defined as 10 consecutive compressions that fail to meet AHA guidelines for depth and rate) and mean time to anaerobic threshold in each manikin.
Effect of Step stool use | 3 years
  The endpoint will be the difference between mean time to ineffective compressions (defined as 10 consecutive compressions that fail to meet AHA guidelines for depth and rate) and mean time to anaerobic threshold in each experimental group.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) Score | 3 years
  Correlation between VAS score and time to ineffective compressions
Physiologic measures and CC quality | 3 years
  Correlation between physiologic measures [anaerobic threshold, Minute oxygen consumption (VO2), Minute carbon dioxide production (VCO2), Oxygen pulse (O2P), Maximal minute ventilation (VE) and Respiratory Exchange Ratio (RER)] and time to ineffective compressions;
Effect of stepstool use on duration of effective compressions. | 3 yrs
• Correlation of subjective reviewer rating and quantitative objective chest compression quality. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Fran Nadel, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Badaki-Makun O, Nadel F, Donoghue A, McBride M, Niles D, Seacrist T, Maltese M, Zhang X, Paridon S, Nadkarni VM. Chest compression quality over time in pediatric resuscitations. Pediatrics. 2013 Mar;131(3):e797-804. doi: 10.1542/peds.2012-1892. Epub 2013 Feb 25. PMID 23439892